CLINICAL TRIAL: NCT03433469
Title: A Phase II Study to Evaluate Neoadjuvant Osimertinib Therapy in Patients With Surgically Resectable, EGFR-Mutant Non-Small Cell Lung Cancer
Brief Title: Osimertinib in Treating Participants With Stage I-IIIA EGFR-mutant Non-small Cell Lung Cancer Before Surgery
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17658; NCI-2018-00019 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-01-25; First posted 2018-02-14 (Actual); Results first posted 2024-01-18 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Stage I Non-Small Cell Lung Cancer; Stage IA Non-Small Cell Lung Cancer; Stage IB Non-Small Cell Lung Cancer; Stage II Non-Small Cell Lung Cancer; Stage IIA Non-Small Cell Lung Cancer; Stage IIB Non-Small Cell Lung Cancer; Stage IIIA Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (osimertinib) (Experimental): Participants receive 80mg osimertinib orally, once a day (PO QD) on days 1-28. Treatment repeats every 28 days for a minimum of 1 cycle prior to surgery in the absence of disease progression or unacceptable toxicity. Investigators will have the option to give a second cycle of study drug prior to surgery if clinically indicated. Depending on the timing of the final scans, patients may ultimately receive up to two weeks additional therapy with study drug beyond end of cycle 1 (or cycle 2) while awaiting surgery. Patients then undergo surgical resection of their cancer. No treatment with the study drug will be given after surgery.
  Interventions: Drug: Osimertinib; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Osimertinib — Given PO (orally)
  Other Names: AZD-9291; Tagrisso
Procedure: Therapeutic Conventional Surgery — Undergo surgery

SUMMARY:
This phase II trial studies how well osimertinib works in treating participants with stage I-IIIA Epithelial Growth Factor Receptor (EGFR) -mutant non-small cell lung cancer before surgery. Osimertinib may stop the growth of tumor cells by blocking mutant EGFR signaling in cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of osimertinib as neoadjuvant therapy in patients with surgically resectable EGFR-mutant non-small cell lung cancer (NSCLC).

SECONDARY OBJECTIVES:

I. To evaluate the safety of osimertinib given as neoadjuvant therapy in early stage EGFR-mutant NSCLC participants.

II. To evaluate whether neoadjuvant osimertinib treatment increases the frequency of tumors that are unresectable due to adverse events or disease progression.

III. To evaluate secondary measures of clinical efficacy in early stage EGFR-mutant NSCLC patients treated with osimertinib induction therapy.

TERTIARY OBJECTIVES:

I. To evaluate long-term measures of efficacy in patients treated with osimertinib neoadjuvant therapy.

II. To explore tissue and cell-free biomarkers that may be predictive of response or primary resistance to osimertinib neoadjuvant therapy.

OUTLINE:

Participants receive osimertinib orally (PO) once daily (QD) on days 1-28. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo surgical resection of their cancer.

After completion of study treatment, participants are followed up at 30 days then every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Males and females >=18 years of age
* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC), performed on a biopsy that occurred within the last 90 days. This biopsy can be deferred if the procedure is deemed to represent an unacceptable safety risk to the patient by the Principal Investigator and as long as the patient has a prior biopsy showing non-small cell lung cancer.
* Documented activating EGFR mutation (Exon 19 deletion, T790M, or L858R) on tumor samples by Clinical Laboratory Clinical Laboratory Improvement Amendments (CLIA)-approved test
* Patients treated with osimertinib or another EGFR tyrosine kinase inhibitors (TKI) (including erlotinib, afatinib, gefitinib, & rocelitinib) are eligible if they received no more than 28 days of treatment, and if there is no evidence of grade 2 or greater treatment adverse events possibly related to treatment with the EGFR TKI.
* Positron emission tomography (PET)-computed tomography (CT) within the last 60 days showing radiographic stage I to IIIa lung cancer (mediastinal staging biopsy is allowed but not required)
* Brain magnetic resonance imaging (MRI) (or CT if contraindication to MRI) within the last 60 days showing no evidence of metastatic disease
* Documentation that the patient is a candidate for surgical resection of their lung cancer by an American Board of Thoracic Surgery certified surgeon
* The patient must have a tumor size >=1 centimeter (cm) in its longest diameter.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0-1
* Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of starting study treatment, with the exception of alopecia and grade 2 prior platinumtherapy-related neuropathy is allowed
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN)
* Bilirubin =< 1.5 x ULN, (Patients with documented Gilbert's syndrome and conjugated bilirubin within the normal range may be allowed into the study; in this event, it will be documented that the patient was eligible based on conjugated bilirubin levels)
* Potassium and magnesium within normal range, patients may receive supplements to meet this requirement
* Leukocytes > 3,000/microliter (mcL)
* Hemoglobin >= 9 g/dL, with no blood transfusions in the 28 days prior to study entry
* Absolute neutrophil count > 1,500/mcL
* Platelets > 100,000/mcL
* Creatinine Clearance (CrCl) > 50 mL/min for patients with serum creatinine (SCr) > 1.5 x upper limit of normal (ULN)
* Ability to swallow oral medications
* Women of childbearing potential (WoCBP) must have a negative serum pregnancy test within 3 days prior to the first dose of study treatment and agree to use highly effective contraception, during the study and for 90 days following the last dose of osimertinib

  * Women of childbearing potential (WoCBP): women between menarche and menopause who have not been permanently or surgically sterilized and are capable of procreation
  * Women NOT of childbearing potential: women who are permanently or surgically sterilized or postmenopausal

    * Permanent sterilization includes hysterectomy and/or bilateral oophorectomy and/or bilateral salpingectomy but excludes bilateral tubal occlusion; tubal occlusion is considered a highly effective method of birth control but does not absolutely exclude possibility of pregnancy; (the term occlusion refers to both occluding and ligating techniques that do not physically remove the oviducts)
  * Women who have undergone tubal occlusion should be managed on trials as if they are of WoCBP (e.g. undergo pregnancy testing etc., as required by the study protocol)
  * Women will be considered postmenopausal if they are amenorrhoeic for 12 months without an alternative medical cause; the following age-specific requirements apply:

    * Women under 50 years old will be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and with luteinizing hormone and follicle-stimulating hormone levels in the postmenopausal range
    * Women over 50 years of age will be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatments
  * Acceptable contraception methods are:

    * Total sexual abstinence (abstinence must be for the total duration of the trial and the follow-up period)
    * Vasectomized sexual partner plus male condom (with participant assurance that partner received post-vasectomy confirmation of azoospermia)
    * Tubal occlusion plus male condom
    * Intra-uterine device - provided coils are copper-banded, plus male condom
    * Intra-uterine system (IUS) levonorgestrel IUS (e.g., Mirena), plus male condom
    * Medroxyprogesterone injections (Depo-Provera) plus male condom
    * Etonogestrel implants (e.g., Implanon, Norplan) plus male condom
    * Normal and low dose combined oral contraceptive pills, plus male condom
    * Norelgestromin / ethinylestradiol transdermal system plus male condom
    * Intravaginal device (e.g., ethinylestradiol and etonogestrel) plus male condom
    * Cerazette (desogestrel) plus male condom (Cerazette is currently the only highly efficacious progesterone based pill)
  * Unacceptable Contraception Methods The following methods are considered not to be highly effective and are therefore not acceptable contraceptive methods:

    * Triphasic combined oral contraceptives
    * All progesterone only pills except, Cerazette
    * All barrier methods, if intended to be used alone
    * Non-copper containing intra-uterine devices
    * Fertility awareness methods
    * Coitus interruptus
* Men with a female partner of childbearing potential must have either had a prior vasectomy agree to use effective contraception as described in the full protocol for at least 14 days prior to administration of the first dose of study treatment, during the study, and for 90 days following the last dose of osimertinib

Exclusion Criteria:

* Leptomeningeal carcinomatosis or other central nervous system (CNS) metastases
* Stage IIIB, or distant metastases (including malignant pleural effusion) identified on PET-CT scan or biopsy (PET abnormalities that are negative for malignancy on biopsy will be considered on a case by case basis
* Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease
* Patients who are known to be serologically positive for human immunodeficiency virus (HIV)
* Active second malignancy, i.e. patient known to have potentially fatal cancer present for which he/she may be (but not necessarily) currently receiving treatment; patients with a history of malignancy that has been completely treated, with no evidence of that cancer currently, are permitted to enroll in the trial provided all chemotherapy for prior malignancy was completed > 12 months prior and/or bone marrow transplant > 2 years prior
* Patients who are currently receiving treatment with contraindicated corrected QT interval (QTc) prolonging medications or potent CYP3A4 inducers, if that treatment cannot be either discontinued or switched to a different medication prior to first day of study treatment. All patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer effects
* Any of the following cardiac abnormalities or history:

  * Mean resting corrected QT interval (QTc) > 470 msec, obtained from 3 electrocardiograms (ECGs), using the screening clinic ECG machine derived QTc value
  * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG e.g. complete left bundle branch block, third degree heart block and second degree heart block
  * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval
* Treatment with prohibited medications (concurrent anticancer therapy including chemotherapy, radiation, hormonal treatment [except corticosteroids and megesterolacetate], or immunotherapy) =< 14 days prior to treatment with osimertinib
* Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator?s opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol, or known active infection including chronic active hepatitis B, hepatitis C and human immunodeficiency virus (HIV); screening for chronic conditions is not required; patients with chronic hepatitis B virus (HBV) with negative HBV viral load on appropriate antiviral therapy will be permitted, if able to continue appropriate antiviral therapy throughout treatment period
* Active tuberculosis
* Signs or symptoms of infection within 2 weeks prior to first day of study
* Therapeutic oral or intravenous (IV) antibiotics within 2 weeks prior to first day of study treatment:

  * Patients receiving prophylactic antibiotics (eg, to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible
* Class II to IV heart failure as defined by the New York Heart Association functional classification system
* Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or left ventricular ejection fraction (LVEF) < 50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate, to be eligible
* Patients who have experienced untreated and/or uncontrolled cardiovascular conditions and/or have symptomatic cardiac dysfunction (unstable angina, congestive heart failure, myocardial infarction within the previous 3 months; coronary angioplasty, or stenting or bypass grafting within the past 6 months; cardiac ventricular arrhythmias requiring medication; any history of second (2nd) or third (3rd) degree atrioventricular conduction defects)
* Females who are pregnant or breastfeeding
* Presence of active gastrointestinal (GI) disease (including GI bleeding or ulceration) or other condition that could affect GI absorption (e.g. malabsorption syndrome, history of biliary tract disease), including refractory nausea or vomiting, or chronic GI disease which may affect absorption or tolerance to oral medications
* History of hypersensitivity to active or inactive excipients of osimertinib or drugs with a similar chemical structure or class to osimertinib
* Involvement in the planning and/or conduct of the study (applies to both investigator staff and/or staff at the study site)
* Participation in another clinical study with an investigational product during the last 2 months or within five half-lives of the compound, whichever is longer
* Uncontrolled medical, psychological, familial, sociological, or geographical conditions that interfere with the patient?s safety, ability to provide informed consent, or ability to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2026-10-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Collin Blakely, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - University of California, Davis, Davis, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blakely CM, Urisman A, Gubens MA, Mulvey CK, Allen GM, Shiboski SC, Rotow JK, Chakrabarti T, Kerr DL, Aredo JV, Bacaltos B, Gee M, Tan L, Jones KD, Devine WP, Doebele RC, Aisner DL, Patil T, Schenk EL, Bivona TG, Riess JW, Coleman M, Kratz JR, Jablons DM. Neoadjuvant Osimertinib for the Treatment of Stage I-IIIA Epidermal Growth Factor Receptor-Mutated Non-Small Cell Lung Cancer: A Phase II Multicenter Study. J Clin Oncol. 2024 Sep 10;42(26):3105-3114. doi: 10.1200/JCO.24.00071. Epub 2024 Jul 19. PMID 39028931

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Osimertinib): Participants receive 80mg osimertinib orally, once a day (PO QD) on days 1-28. Treatment repeats every 28 days for a minimum of 1 cycle prior to surgery in the absence of disease progression or unacceptable toxicity. Investigators will have the option to give a second cycle of study drug prior to surgery if clinically indicated. Depending on the timing of the final scans, participants may ultimately receive up to two weeks additional therapy with study drug beyond end of cycle 1 (or cycle 2) while awaiting surgery. Participants then undergo non-investigational surgical resection of their cancer. No treatment with the study drug will be given after surgery.
Period: Overall Study
Arm/Group | Treatment (Osimertinib)
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Osimertinib)
Number analyzed (Participants) | 27
Age, Customized [Count of Participants; unit: Participants]
  30-39 years old | 1
  40-49 years old | 2
  50-59 years old | 4
  60-69 years old | 8
  70-79 years old | 9
  80-89 years old | 3
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 20
  Male | 6
  Not reported/Unknown/Declined to State | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Major Pathological Response (MPR)
Description: Tumors that exhibit =< 10% viable tumor will meet the criteria for a major pathological response. MPR will be determined in patients who receive at least one dose of study drug and become ineligible for surgery either because of disease progression or adverse event will be deemed not to have achieved MPR. The major pathological response rate will be reported with 95% confidence intervals.
Time Frame: Up to 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Osimertinib)
Number analyzed (Participants) | 27
percentage of participants | 14.8 [5.9 to 32.5]

2. Secondary Outcome: Objective Response Rates (ORR)
Description: The percentage of participants with a best overall response rate of complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD) determined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria and by investigator's assessment will be determined from the time of treatment until surgery. The frequency and percentages of patients with a best ORR of CR, PR, SD, or PD will be determined. The ORR for each response type will be reported with 95% confidence intervals.
Time Frame: Up to 70 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Osimertinib)
Number analyzed (Participants) | 27
percentage of participants
  Complete Response (CR) | 0 [0 to 12.5]
  Partial Response | 51.9 [34 to 69]
  Stable Disease | 44.4 [27.6 to 62.7]
  Progressive Disease | 3.7 [0.2 to 18.3]

3. Secondary Outcome: Mean Disease-free Survival (DFS)
Description: DFS will be calculated as 1+ the number of days from date of surgical resection to documented radiographic relapse/progression or death due to any cause over a period of 60 months. The Kaplan-Meier analysis will be used to calculate the median DFS with 95% confidence interval.
Time Frame: Up to 5 years
Reporting Status: Not Posted

4. Secondary Outcome: Disease-free Survival Rate (DFS)
Description: DFS will be calculated as 1+ the number of days from date of surgical resection to documented radiographic relapse/progression or death due to any cause over a period of 60 months. The 5-year DFS rate will be calculated as the percentage of patients who are disease free at 5 years. This will be calculated using the Kaplan-Meier method
Time Frame: Up to 5 years
Reporting Status: Not Posted

5. Secondary Outcome: Overall Survival (OS)
Description: 5-year OS rate will be calculated using the Kaplan-Meier method . OS will be defined as the 1+ the number of days from surgical resection to death due to any cause over a period of 60 months. The Kaplan-Meier analysis will be used to calculate the median OS with 95% confidence interval.
Time Frame: Up to 5 years
Reporting Status: Not Posted

6. Secondary Outcome: Median Percentage Change in Tumor Burden (Depth of Response)
Description: Depth of response (DpR) will be defined as the percentage change in tumor burden by RECIST criteria at best response versus baseline imaging. DpR will be summarized using descriptive statistics.
Time Frame: Up to 1 year
Measure: Median (95% Confidence Interval); unit: percent change
Arm/Group | Treatment (Osimertinib)
Number analyzed (Participants) | 27
percent change | -32 [-40 to -18]

7. Secondary Outcome: Pathologic Complete Response Rate (pCR)
Description: The pCR is defined as absence of (0%) viable tumor present histologically in the resected tumor specimen
Time Frame: Up to 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Osimertinib)
Number analyzed (Participants) | 27
percentage of participants | 0 [0 to 12.5]

8. Secondary Outcome: Percentage of Participants With of Treatment-related Adverse Events (AEs)
Description: The percentage of participants with treatment-related adverse events will be reported. Adverse events will be classified according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: Up to 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Osimertinib)
Number analyzed (Participants) | 27
percentage of participants | 100

9. Secondary Outcome: Percentage of Participants Unable to Undergo Surgical Resection
Description: Rate of conversion from operable to non-operative will be recorded as rate of patients initially assessed as surgically resectable, who are subsequently unable to undergo surgical resection due to either treatment-related adverse events (AEs) or disease progression.
Time Frame: Up to 70 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Osimertinib)
Number analyzed (Participants) | 27
percentage of participants | 11.1 [3.9 to 28.1]

10. Secondary Outcome: Percentage of Surgical Complications
Description: Rate of surgical complications occurring prior to the end of treatment visit will be reported
Time Frame: Up to 1 year
Population: Three participants were deemed not to be surgical candidates by the investigator at the time of surgery following treatment and were excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Osimertinib)
Number analyzed (Participants) | 24
percentage of participants | 62.5 [42.7 to 78.8]

ADVERSE EVENTS:
Time Frame: Up to 1 year
Description: Collection for long term survival up to 5 years is still ongoing.
Arm/Group | Treatment (Osimertinib)
All-Cause Mortality (participants affected / at risk) | 4/27
Serious Adverse Events (participants affected / at risk) | 3/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Osimertinib) (N=27)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Osimertinib) (N=27)
Diarrhea (Gastrointestinal disorders) | 13 (16)
Nausea (Gastrointestinal disorders) | 7 (7)
Dry mouth (Gastrointestinal disorders) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2)
Dry Skin (Skin and subcutaneous tissue disorders) | 5 (5)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 3 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Fatigue (General disorders) | 8 (8)
Fever (General disorders) | 2 (2)
Neutrophil count decreased (Investigations) | 3 (5)
Alanine aminotransferase increased (Investigations) | 2 (5)
Aspartate aminotransferase increased (Investigations) | 2 (4)
Platelet count decreased (Investigations) | 2 (2)
White blood cell decreased (Investigations) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 3 (4)
Headache (Nervous system disorders) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2)
Blurred vision (Eye disorders) | 3 (3)
Dry Eye (Eye disorders) | 2 (2)
Paronychia (Infections and infestations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (4)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/69/NCT03433469/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-15): https://cdn.clinicaltrials.gov/large-docs/69/NCT03433469/ICF_001.pdf